CLINICAL TRIAL: NCT03277391
Title: Serratus Anterior Plane Block: Post-operative Analgesia Technique in Video-assisted Thoracic Surgery. Efficacy Pilot Study and Population Pharmacokinetic Analysis
Brief Title: Serratus Anterior Plane Block: Post-operative Analgesia in Video-assisted Thoracic Surgery
Acronym: Serrathos
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Paul Gruson, Principal investigator, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P2017/170
Record Dates: First submitted 2017-08-25; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Regional Anesthesia; Thoracic Surgery; Post-operative Pain; Post-operative Chronic Pain; Pharmacokinetic Analysis; Serratus Anterior Plane Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant
Masking Description: Random attribution by computer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus anterior plane block (Active Comparator): Deep serratus anterior plane block
  Interventions: Procedure: Serratus anterior plane block; Device: patient-controlled analgesia
- patient-controlled analgesia (Active Comparator): patient-controlled analgesia: pump containing morphine (1mg/ml) and dehydrobenzperidol (50 mcg/ml).
  Interventions: Device: patient-controlled analgesia

INTERVENTIONS:
Procedure: Serratus anterior plane block — SPB realized under ultrasound guidance. Infiltration of local anesthetic (bolus then infusion through a multi-holed catheter) is realized under the serratus anterior muscle at a level situated around the 5th to 6th intercostal space on the anterior axillary lign, in order to anesthetize the cutaneous lateral branches of the intercostal nerves, with a first ropivacaine 0,375% bolus (0,4ml/kg), followed by an infusion of ropivacaine 0,2% at a 10ml/hr rate, through a multi-holed catheter, for a duration of 24 hours.
  Other Names: Deep serratus anterior plane block; SPB
  Arms: Serratus anterior plane block
Device: patient-controlled analgesia — Each patient controls his analgesia with an IV bolus of 2mg of morphine every 10 minutes if needed, with a maximum of 20mg every 4 hours.
  Other Names: PCA morphine dehydrobenzperidol

SUMMARY:
The objective of the study is to compare the efficacy of the Serratus Anterior Plane block (SPB) realised in its deep plane, with a multi-holed catheter in place for twenty four hours, to a standard intravenous analgesia for small videoassisted thoracic surgery interventions. The objective is also to evaluate the resorption rate of local anesthetic at this level, and make a population pharmacokinetic analysis.

DETAILED DESCRIPTION:
In this study, 20 patients will be randomly assigned to one of two groups: ten patients will have a Serratus anterior plane block (SPB), with a first ropivacaine 0,375% bolus (0,4ml/kg), followed by an infusion of ropivacaine 0,2% at a 10ml/hr rate, through a multi-holed catheter located under the serratus anterior muscle, for a duration of 24 hours. The other group will have a standard intravenous analgesia with a PCA morphine-dehydrobenzperidol pump. Anesthesia protocol will be standardized. Except the infusion of ropivacaine for the SPB, per operative anesthesia and post operative analgesia will be the same for every usual patients.

The investigators will evaluate post operative pain based on the visual analog scale, 24 hours morphine consumption, sensitivity of concerned territory. The investigators will also evaluate post operative chronic pain by assessing pain two months post operatively, completing two questionnaires of neuropathic pain: DN4 and QDSA short form.

Finally, ropivacaine blood concentrations will be dosed by multiple blood samples taken over 24 hours after realizing the SPB, in order to make a population pharmacokinetic analysis, and evaluate the degree of ropivacaine resorption at this level.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists physic status 1, 2 and 3 who require surgical video-assisted thoracoscopy or video assisted thoracic surgery without mini-thoracotomy

1. Lung pathologies:

   * biopsies
   * symphysis, pleurectomy
   * emphysema bullae resection
2. pleural pathologies:

   * biopsies
   * collections, intra pleural effusion
3. mediastinal pathologies:

   * adenopathy staging
   * cysts
   * sympathectomy T2-T5
   * vagotomy
   * splanchnicectomy

Exclusion Criteria:

1. refusal
2. allergy to local anesthetic - contra-indication to the use of ropivacaine
3. pregnancy
4. liver failure
5. severe kidney disease (GFR < 15ml/min)
6. chronic intake of opioids
7. neurological or psychiatric disorders interfering with pain assessment
8. severe and morbid obesity (BMI > 35)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption (mg) | 24 hours
  Consumption of intravenous morphine

SECONDARY OUTCOMES:
Pain score | 24 hours
  Visual Analog Score: assess pain on surgical site
Post operative nausea | 24 hours
  Presence or absence of nausea
Post operative vomiting | 24hrs
  Presence or absence of vomiting
Sensitivity of SPB zone | 24 hours
  Cold (ether) applied on the skin of the operated hemithorax
Post operative chronic pain | 2 months
  Two months after surgery: QDSA-sf (short form of Questionnaire de douleur de Saint-Antoine)
Post operative chronic pain | 2 months
  Two months after surgery: DN4 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Luc Van Obbergh, Principal Investigator — Anesthesiology chief
Locations (1):
- Hopital Erasme, Anderlecht, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor R, Massey S, Stuart-Smith K. Postoperative analgesia in video-assisted thoracoscopy: the role of intercostal blockade. J Cardiothorac Vasc Anesth. 2004 Jun;18(3):317-21. doi: 10.1053/j.jvca.2004.03.012. PMID 15232812
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Font MC, Navarro-Martinez J, Nadal SB, Munoz CG, Galiana-Ivars M, Montero PC. Continuous Analgesia Using a Multi-Holed Catheter in Serratus Plane for Thoracic Surgery. Pain Physician. 2016 May;19(4):E684-5. No abstract available. PMID 27228541
- [Background] Madabushi R, Tewari S, Gautam SK, Agarwal A, Agarwal A. Serratus anterior plane block: a new analgesic technique for post-thoracotomy pain. Pain Physician. 2015 May-Jun;18(3):E421-4. PMID 26000690
- [Background] Broseta AM, Errando C, De Andres J, Diaz-Cambronero O, Ortega-Monzo J. Serratus plane block: the regional analgesia technique for thoracoscopy? Anaesthesia. 2015 Nov;70(11):1329-30. doi: 10.1111/anae.13263. No abstract available. PMID 26449303
- [Background] Cruccu G, Sommer C, Anand P, Attal N, Baron R, Garcia-Larrea L, Haanpaa M, Jensen TS, Serra J, Treede RD. EFNS guidelines on neuropathic pain assessment: revised 2009. Eur J Neurol. 2010 Aug;17(8):1010-8. doi: 10.1111/j.1468-1331.2010.02969.x. Epub 2010 Mar 8. PMID 20298428
- [Background] Dworkin RH, Turk DC, Trudeau JJ, Benson C, Biondi DM, Katz NP, Kim M. Validation of the Short-form McGill Pain Questionnaire-2 (SF-MPQ-2) in acute low back pain. J Pain. 2015 Apr;16(4):357-66. doi: 10.1016/j.jpain.2015.01.012. Epub 2015 Jan 29. PMID 25640290
- [Background] Kopacz DJ, Emanuelsson BM, Thompson GE, Carpenter RL, Stephenson CA. Pharmacokinetics of ropivacaine and bupivacaine for bilateral intercostal blockade in healthy male volunteers. Anesthesiology. 1994 Nov;81(5):1139-48. doi: 10.1097/00000542-199411000-00007. PMID 7978472
- [Background] Scott DB, Lee A, Fagan D, Bowler GM, Bloomfield P, Lundh R. Acute toxicity of ropivacaine compared with that of bupivacaine. Anesth Analg. 1989 Nov;69(5):563-9. PMID 2679230
- [Result] Joshi GP, Bonnet F, Shah R, Wilkinson RC, Camu F, Fischer B, Neugebauer EA, Rawal N, Schug SA, Simanski C, Kehlet H. A systematic review of randomized trials evaluating regional techniques for postthoracotomy analgesia. Anesth Analg. 2008 Sep;107(3):1026-40. doi: 10.1213/01.ane.0000333274.63501.ff. PMID 18713924